CLINICAL TRIAL: NCT01943045
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Multiple Center Study to Evaluate the Safety, Tolerability, and Activity of NGM282 Administered for 28 Days to Patients With Type 2 Diabetes Mellitus
Brief Title: Phase 2 Study of NGM282 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Collaborators: NGM Biopharmaceuticals Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0102
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NGM282 Dose 1 (Experimental): NGM Dose 1
  Interventions: Biological: NGM282
- NGM282 Dose 2 (Experimental): NGM Dose 2
  Interventions: Biological: NGM282
- NGM282 Dose 3 (Experimental): NGM Dose 3
  Interventions: Biological: NGM282
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NGM282
  Arms: NGM282 Dose 1; NGM282 Dose 2; NGM282 Dose 3
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and activity of NGM282 in patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 70 years of age, inclusive
* BMI range of 24-40 kg/m2, inclusive
* No active coronary artery disease
* Resting heart rate in the range of 40-100 bpm

Exclusion Criteria:

* Diagnosis of Type 1 diabetes
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma Glucose | 28 days

SECONDARY OUTCOMES:
HbA1c | 28 days
Lipids | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Alex M DePaoli, MD, Study Director — NGM Biopharmaceuticals, Inc
Locations (9):
- Australia (3):
  - NGM Clinical Study Site 6103, Melbourne, Victoria
  - NGM Clinical Study Site 6104, Melbourne, Victoria
  - NGM Clinical Study Site 6101, Perth, Western Australia
- New Zealand (6):
  - NGM Clinical Study Site 6403, Auckland
  - NGM Clinical Study Site 6405, Auckland
  - NGM Clinical Study Site 6401, Christchurch
  - NGM Clinical Study Site 6406, Dunedin
  - NGM Clinical Study Site 6404, Tauranga
  - NGM Clinical Study Site 6402, Wellington

REFERENCES:
- [Derived] DePaoli AM, Zhou M, Kaplan DD, Hunt SC, Adams TD, Learned RM, Tian H, Ling L. FGF19 Analog as a Surgical Factor Mimetic That Contributes to Metabolic Effects Beyond Glucose Homeostasis. Diabetes. 2019 Jun;68(6):1315-1328. doi: 10.2337/db18-1305. Epub 2019 Mar 12. PMID 30862680
- See also: Related Info — http://ngmbio.com/